CLINICAL TRIAL: NCT03458676
Title: Radiologic Pathologic Correlation of Advanced MR Imaging to Guide the Biopsy of Cerebral Malignancies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011-0370; NCI-2018-00924 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2018-03-02; First posted 2018-03-08 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Brain Lesion
Keywords: Advanced magnetic resonance imaging; AMRI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Advanced MR Imaging (AMRI) Scan (Experimental): AMRI scan performed within 2 weeks before standard of care brain surgery.
  During the surgery, neurosurgeon(s) use the information collected from the AMRI to decide what area of the brain tumor will be biopsied.
  Interventions: Procedure: Advanced Magnetic Resonance Imaging Scan; Procedure: Standard of Care Brain Biopsy and Tumor Removal

INTERVENTIONS:
Procedure: Advanced Magnetic Resonance Imaging Scan — AMRI scan performed within 2 weeks before standard of care brain biopsy and tumor removal surgery.
  AMRI scan should take less than 1 hour to complete
  Other Names: AMRI
Procedure: Standard of Care Brain Biopsy and Tumor Removal — During the surgery, the neurosurgeon(s) uses the information collected from the AMRI to decide what area of the brain tumor will be biopsied.
  Biopsies from up to 5 locations taken before the tumor is surgically removed.

SUMMARY:
The goal of this clinical research study is to learn if using advanced magnetic resonance imaging (AMRI) will improve the targeting of brain tumor needle biopsies compared to the standard targeting techniques. Researchers also want to learn how the results of the images and biopsies compare to each other to try to improve the way researchers and radiologists use AMRI images.

This is an investigational study. The perfusion scan is not FDA approved or commercially available. It is currently only being used in research.

There will be no cost to you for the advanced MRI, additional anesthesia, special pathology stains, and/or gene testing for this study.

Up to 50 patients will take part in this study. All will be enrolled at MD Anderson.

DETAILED DESCRIPTION:
Participant is being asked to take part in this study because participant has a lesion in participant's brain which is suspected or proven to be a tumor and participant has been scheduled for surgery to remove it.

Some parts of brain tumors are more aggressive than other parts. A needle biopsy only gets a small part of the brain tumor cells. Doctors (neurosurgeons) want to get a biopsy sample from the most aggressive part of the tumor. Researchers think that AMRI techniques may help to better target the most aggressive part of the tumor for the needle biopsy.

AMRI Scan:

In addition to the images that will be taken as part of participant's standard of care surgery preparation, participant will have an AMRI scan performed. The AMRI has several parts. There are 2 perfusion scans that use a contrast dye to look at small blood vessels. There is a spectroscopy scan to looks at the chemical make-up of the tumor. There is also a diffusion scan to look at how water moves in the tumor and can see the white matter that connects both sides of brain parts. The AMRI scans are performed in the same way as normal MRI scans and in the same scanner. They can be noisy, but do not feel any different than standard MRI exams.

In most cases, the AMRI should take less than 1 hour to complete and will be performed within 2 weeks before participant's standard of care surgery.

Surgery During the surgery, the neurosurgeon(s) will use the information collected from the AMRI to decide what area of the brain tumor will be biopsied. The biopsies are only from areas that would normally be cut out during surgery and will not change the way the surgery is done even if participant chooses not to take part in this study. Biopsies (from up to 5 locations, each smaller than participant's thumbnail) will be taken before the tumor is surgically removed. The tumor tissue samples from the biopsies will be tested to learn more about the tumor and optionally the DNA inside(the genetic material of cells - this procedure is described in the optional procedures section below).

After the surgery is over, participant will continue to have participant's standard of care follow-up appointments in the neurosurgery clinic.

Length of Study After the biopsy is complete, your active participation on this study will be over. Participant's medical records will continue to be reviewed for up to an additional 5 years.

Follow-Up Medical Record Review:

After participant's active participation on this study is over, participant's medical record will be reviewed to learn how participant is doing, what other treatments participant may have had and how they worked, if participant had any new brain problems or if the tumor came back. Researchers will review and record information from participant's medical records for up to 5 years after participant's active participation on this study is over.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is >18 years old, agrees to participate in the clinical study and to complete all required visits and evaluations. The pediatric population has a different disease profile from the glioma patients we hope to recruit. To reduce heterogeneity in the patient population we will not consider patients younger than 18 for this study.
2. Patient is a candidate for cerebral tumor resection with lesion suspected to be or previously biopsy proven to be a primary brain tumor.
3. Patient is able to understand and give consent to participation in the study.
4. Patient agrees to undergo, prior to the procedure, magnetic resonance imaging (MRI, within 14 days and preferably with 3 days of the planned procedure) with perfusion, diffusion and spectroscopic imaging. As per study chair's judgement, imaging outside this time window will also be permitted, for suspected slow growing tumors.

Exclusion Criteria:

1. The patient is found to have unfavorable anatomy to indicate that stereotactic biopsy could not be safely performed.
2. Renal failure as evidenced by a GFR of less than 30 mL/min/1.73m2 for gadolinium based imaging, for iodinated contrast agent we will use the more strict cut-off of 45 mL/min/1.73m2 (Davenport, 2020, Radiology: Use of IV Iodinated contrast media in patients with Kidney Disease: Consensus statement from the ACR and the National Kidney Foundation). This differentiation reflects the different risk profiles of these agents, and are conservative when compared to our clinical practice. In the absence of eGFR lab result, patient is not excluded in the absence of remarkable pathological renal history as confirmed by and in the discretion of the PI. As per current departmental guidelines, late-generation gadolinium contrast agents (such as gadobutrol and gadopiclenol), can still be administered safely in the setting of low renal function, provided clinical risk-benefit is maintained.
3. Pacemakers, electronic stimulation, metallic foreign bodies and devices and/or other conditions that are not MR safe, which include but are not limited to:

   * electronically, magnetically, and mechanically activated implants
   * ferromagnetic or electronically operated active devices like automatic cardioverter defibrillators and cardiac pacemakers
   * metallic splinters in the eye
   * ferromagnetic hemostatic clips in the central nervous system (CNS) or body
   * cochlear implants
   * other pacemakers, e.g., for the carotid sinus
   * insulin pumps and nerve stimulators
   * non-MR safe lead wires
   * prosthetic heart valves (if dehiscence is suspected)
   * non-ferromagnetic stapedial implants
   * pregnancy
   * claustrophobia that does not readily respond to oral medication 4. Allergy to relevant imaging contrast agents, includes allergies to iodine or gadolinium-based contrast agents (if one class of agents is contra-indicated, then imaging with the other can still proceed).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2012-09-06 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of the Accuracy of the Pathological Grades of Tumor Observed at the Biopsy Locations Identified Using Conventional Versus Advanced Imaging | 2 weeks
  Researchers wish to determine if the accuracy of the pathological grade observed at the biopsy sites identified by advanced imaging is higher than the grades observed at the biopsy sites identified by conventional imaging.
Target Sample Grading | 2 weeks
  The quantitative pathology markers compared between the conventional and advanced target specimens.

CONTACTS AND LOCATIONS:
Overall Officials: Dawid Schellingerhout, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org